CLINICAL TRIAL: NCT06275165
Title: The Effects of Acupressure on Improving Postoperative Gastrointestinal Symptom Distress in Esophageal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHEN, CHIA-CHEN (Other)
Responsible Party: Sponsor-Investigator, CHEN, CHIA-CHEN, Principal Investigator, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202301754B0
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Esophageal Cancer; Gastrointestinal Dysfunction
Keywords: gastrointestinal symptom distress; acupressure
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Participants were divided into an experimental group and a control group. experimental group: received acupressure for 5 days in addition to regular care.
  control group: received regular postoperative care.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure (Experimental): Participants received routine care and acupressure.
  Interventions: Other: acupressure
- no intervision (No Intervention): received routine care

INTERVENTIONS:
Other: acupressure — In the experimental group, routine nursing care and acupressure (Neiguan and Zusanli points) were performed from the 1st to the 5th day after the postoperative transfer from the ward to the hospital room. Twice a day, 3 minutes each time, 12 minutes in total.
  Arms: acupressure

SUMMARY:
This study is a quasi-experimental design clinical trial with the primary objective of comparing the health status of patients with esophageal cancer. Participants were divided into an experimental group and a control group. Patients in the experimental group received routine care and acupressure for 5 consecutive days starting from the day after entering the ward after esophageal cancer surgery, in the control group, participants received routine care, and Participants were assessed on the Gastrointestinal Symptom Distress Scale at the end of the intervention. The aim of this study was to verify the effectiveness of acupressure in improving of gastrointestinal symptoms distress after esophageal cancer surgery.

DETAILED DESCRIPTION:
Esophageal cancer is one of the common and highly fatal malignant tumors, and its incidence rate is increasing every year, and most of them are in the middle and advanced stages when diagnosed. Surgery is the standard treatment for the eradication of esophageal cancer, which can effectively reduce the mortality rate and improve the survival rate, but the patients often experience gastrointestinal discomfort after surgery, which impedes the intake of nutrients and the body's recovery. The purpose of this study was to investigate the effectiveness of acupressure in improving the postoperative gastrointestinal discomfort in patients with esophageal cancer. An experimental study design was adopted, and patients were assigned to the experimental group and the control group in a time-divided manner. The experimental group was assigned to the experimental group and the control group in a time-separated manner. The experimental group received regular care from the first day to the fifth day after the patients were transferred from the intensive care unit to the hospital ward after the surgery, and they received acupressure at the Neiguan point of the upper limbs and the four acupoints of the foot Sanli of the lower limbs twice a day for 3 minutes each, for a total of 12 minutes; while the control group received regular care in the first day of the study. In this study, the gastrointestinal symptoms of the experimental group before and after acupressure were collected and compared with those of the control group, in order to verify the effectiveness of acupressure in improving gastrointestinal symptoms during postoperative nutritional support for jejunostomy.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized men and women who agree to participate in this study
* Patients diagnosed with esophageal cancer based on pathological tissue section results
* Nutritional support through jejunostomy in post esophagectomy patients
* A sufficient level of education to understand study procedures and be able to communicate with site personnel

Exclusion Criteria:

* Pregnant or lactating women
* Diagnosed and treated for peripheral vascular disease within 3 months prior to surgery.
* Those with unstable vital signs and septicemia infection after surgery.
* Those who are suffering from blood diseases with abnormal coagulation function, or Currently taking anticoagulant drugs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in gastrointestinal symptom distress Scale at study day 5(end day) | Baseline and study day 5
  The Gastrointestinal Symptom Distress Scale is a validated self-report tool that assesses 10 gastrointestinal symptoms that patients with esophageal cancer may face after surgery. The 10-question questionnaire measures the self-perceived severity of nausea, vomiting, satiety, bloating, abdominal cramps, acid reflux, chest tightness, heart burn, diarrhea, and constipation, as well as the degree of interference with life. Using an 11-point Likert scale, 0 points (never happened), 1 point (very slight/very slight interference), 10 points (very severe/extreme interference), and the total score of the scale is 0-100 points.
  The higher the measured score, the more severe the gastrointestinal discomfort symptoms are and the more they interfere with life.
  The Gastrointestinal Symptom Distress Scale was subjected to an expert validity review, using the CVI (content validity index) calculation method, and the score was above 0.80.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chen Chen, Principal Investigator — Chang Gung Memorail Hospital
Locations (1):
- Chang Gung Memotial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No